CLINICAL TRIAL: NCT01520870
Title: Phase II Pilot, Prospective, Open Label, Multicenter CT, to Evaluate the Safety and Efficacy of PF299804, a Pan-HER Irreversible Inhibitor, in Patients With Recurrent Glioblastoma With EGFR Amplification or Presence of EGFRvIII Mutation
Brief Title: Safety and Efficacy of PF-299804 (Dacomitinib), a Pan-HER Irreversible Inhibitor, in Patients With Recurrent Glioblastoma With EGFR Amplification or Presence of EGFRvIII Mutation. A Phase II CT.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEINO 11
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Glioblastoma; Brain Tumor, Recurrent
Keywords: Dacomitinib; PF-299804; Glioblastoma, Recurrent; EGFR
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Recurrence | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-299804 (Dacomitinib) (Experimental): Dacomitinib will be administered orally at a dose of 45 mg/day, until disease progression, unacceptable adverse side effects or study end. Patients at first recurrence will be enrolled onto 1 of 2 cohorts that will be recruited and analysed independently. Cohort A will include patients who have EGFRvIII mutations. Cohort B will include patients who have EGFR gene amplification but no EGFRvIII mutations.
  Interventions: Drug: PF-299804 (Dacomitinib)

INTERVENTIONS:
Drug: PF-299804 (Dacomitinib) — Dacomitinib will be administered orally at a dose of 45 mg/day, until disease progression, unacceptable adverse side effects or study end.

SUMMARY:
This multicenter, 2-stage, open-label, phase II trial aims to assess the efficacy and safety of dacomitinib in adult patients with recurrent Glioblastoma (GBM) with EGFR gene amplification and/or EGFRvIII mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign the informed consent approved by the Ethic Committee.
2. Men or women aged greater than or equal to 18.
3. Patients with grade IV malignant glioma according to WHO classification (glioblastoma) in first relapse with histologically confirmed diagnosis by the central laboratory. Patients with previous low-grade glioma or anaplastic glioma (anaplastic astrocytoma or anaplastic oligodendroglioma), are not eligible, even if histological assessment demonstrates transformation to GBM.
4. Patients in first relapse (or progression) to chemo-radiotherapy and temozolomide-based chemotherapy (Stupp4 scheme).
5. All patients must have EGFR gene amplification by in situ hybridization fluorescent (FISH) and / or EGFRvIII mutation by PCR in tumor samples made by the central laboratory (Laboratory of Neuropathology. Hospital Universitario 12 de Octubre).
6. For all study cohorts, patients must be at least 15 unstained slides or a block of paraffin-embedded tissue available from a previous biopsy or surgery (archived tumor samples previously).
7. All patients must show progressive disease of the brain MRI is as defined in the Criteria RANO.
8. Interval of at least one week between prior intra-cranial biopsy, healed properly, and inclusion.
9. Interval of at least 12 weeks between prior radiotherapy and inclusion, unless: a) histopathologic confirmation of recurrent tumor, or b) MR recurrence outside the radiation field.
10. Patients must have recovered from previous therapy: 28 days from the completionof any investigational drug and / or the termination of any cytotoxic therapy.
11. ECOG performance status less than or equal to 2.
12. Stable or decreasing doses of corticosteroids during the five days prior to inclusion in the study.
13. Adequate bone marrow reserve, hematocrit greater than or equal to 29%, WBC> 3000 / mcl,ANC greater than or equal to 1,500 cells / ul, platelets greater than or equal a100.000 cells / ul.
14. Adequate hepatic function: bilirubin less than or equal to 1.5 times ULN, AST (SGOT) less than or equal to 2.5 x ULN.
15. Creatinine within the center ULN or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above the center ULN.
16. The patients in whom resection was made in the first tumor recurrence are eligible in the following cases:

    * There is adequate recovery from surgery.
    * There must be measurable or evaluable disease after surgery. For an adequate Radiological evaluation of residual disease, MRI must be completed within 72 hours after surgery or 4 weeks after surgery.
17. The effects of PF-00299804 in human foetal development are unknown. For this reason, women of childbearing potential and men must agree to use effective contraception (hormonal control method, barrier, abstinence or surgical sterilization) before inclusion in the study, during participating in the study and at least 3 months after treatment has ended the trial. The definition of an effective contraceptive method is based on the criterion of the principal investigator or designee. In case of a woman become pregnant or there is suspicion that she is pregnant while participating in this study, the trial physician must inform immediately. All women of childbearing potential must have a negative pregnancy test (serum / urine) in the 2 weeks before the start of treatment. NOTE: Patients who have received treatment based on the scheme Stupp (Chemoradiotherapy with temozolomide followed by temozolomide sequential) are eligible in the trial, even if other drugs have been added to this scheme. It is excluded from this, those patients who have been treated with EGFR inhibitors for obvious reasons. However, those patients who have received Stupp scheme + other drugs like bevacizumab and cilengitide, remain eligible.

Exclusion Criteria:

1. Presence of extra-cranial metastatic disease.
2. Concomitant treatment with other investigational drugs.
3. Prior treatment with an investigational drug/s known or are suspected to be active by the action of any component of the EGFR tyrosine kinase.
4. Surgery of any kind (does not include diagnostic procedures such as minor lymph node biopsy) in the 2 weeks prior to baseline assessments of the disease, or presence of side effects of previous procedures.
5. Presence of any clinically significant gastrointestinal abnormality that can affect oral administration, transit or absorption of study drug, such as the inability to take medication by mouth as tablets.
6. Presence of any psychiatric or cognitive disorder that limits the understanding or the signature of informed consent and / or jeopardize the fulfillment of the requirements of this protocol.
7. Significant or uncontrolled cardiovascular disease, including:

   * Myocardial infarction within the previous 12 months
   * Uncontrolled angina within the previos 6 months
   * Congestive heart failure in the previous 6 months
   * Known or suspected congenital long QT syndrome
   * History of clinically significant ventricular arrhythmias of any type (as ventricular tachycardia, ventricular fibrillation or torsades de pointes)
   * QTc prolongation on electrocardiogram prior to entry (> 470 msec)
   * History of second or third grade heart block (these patients may be eligible if you currently have a pacemaker)
   * Heart rate < 50/minute in the baseline electrocardiogram
   * Uncontrolled hypertension.
8. Any patient with a history of significant cardiovascular disease, even though is currently controlled, or presents signs or symptoms suggestive of impaired left ventricular function at discretion of the investigator,should have an evaluation of LVEF in these circumstances. If the result is under the center lower limit normal or lower than 50%, the patient would not be eligible.
9. History of any cancer, except for the following circumstances:

   * Patients with a history of other malignancies are eligible if they have been free of disease for at least the last 3 years, and at the discretion of the investigator, there is low risk of disease recurrence.
   * Patients with the following cancers are eligible even if they are diagnosed and treated in the last 3 years: carcinoma in situ of the cervix and basal cell or basal cell skin carcinoma. Patients are ineligible if there is evidence of any neoplastic disease that required therapy other than surgery in the past 3 years.
10. Prior stereotactic radiotherapy or brachytherapy.
11. Intratumoral treatment with CCNU in recurrent tumor surgery (second surgery). NOTE: Patients treated with intratumoral CCNU (or what is the same (intratumor carmustine or Gliadel®), in the first intervention can participate in the study.
12. Presence of leptomeningeal dissemination.
13. Pregnant or breastfeeding. Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects of PF-00299804 is unknown. Because there is an unknown risk of potential adverse effects in infants, secondary to maternal treatment with PF-00299804, breastfeeding should be discontinued if mother is treated with PF-00299804.
14. Patients positive for HIV being treated with antiretroviral combination therapy. These patients are not eligible due to potential pharmacokinetic interactions with PF-00299804. Additionally, these subjects have an increased risk of lethal infections when treated with marrow-suppressive therapy. HIV-positive patients not on antiretroviral combination therapy, are eligible if the disease is controlled at the discretion of the investigator.
15. History of allergic reactions attributed to drugs with similar chemical or biological composition than PF-00299804.
16. Another acute or chronic serious medical condition, uncontrolled intercurrent illness or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of test results and that,investigator's discretion, make the patient inappropriate for entry into this trial. Uncontrolled intercurrent illness including, but are not limited to, ongoing or active infection or psychiatric illness / social situations that limit the compliance of study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2015-04 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sepúlveda, MD, Principal Investigator — Hospital 12 de Octubre
Locations (12):
- Spain (12):
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Barcelona
  - Institut Català D'Oncologia L'Hospitalet (Ico), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario A Coruña, A Coruña, Coruña (A)
  - Hospital Del Mar, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Complejo Hospitalario Regional Virgen de Las Nieves, Granada
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Y Politécnico La Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single-arm study. All patients received the same treatment: Dacomitinib 45 mg/day.
  To obtain a balanced population patients were enrolled in two cohorts depending on their EGFR mutational status. However, most endpoints and baseline characteristics are only analyzed for the full set population, as this was pre-especified per protocol and the interest of the study.
Pre-assignment Details: Patients with first recurrence were enrolled in 2 cohorts. Cohort A included patients with EGFR gene amplification without EGFRvIII mutation. Cohort B included patients with EGFR gene amplification and EGFRvIII mutation.
  All patients received Dacomitinib (45 mg/day) orally until disease progression/unacceptable adverse events (AEs)
Period: Overall Study
Arm/Group | PF-299804 (Dacomitinib)
Started | 49
Completed | 47
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 49
MGMT methylation status [Count of Participants; unit: Participants] — O6-Methylguanine-DNA Methyltransferase (MGMT) is a DNA repair enzyme that removes alkyl adducts from the O6 position of guanine.
  Methylation of the MGMT promoter has been reported in several tumor types.
  Participants
    MGMT methylated | 10
    MGMT non-methylated | 17
    not determined | 22
IDH1/2 mutational status [Count of Participants; unit: Participants] — Mutations in isocitrate dehydrogenase (IDH) 1 and 2 occur in the vast majority of low grade gliomas and secondary high grade gliomas. These mutations change the function of the enzymes, causing increased methylation in gliomas. Gliomas with mutated IDH1 and IDH2 have improved prognosis compared to gliomas with wild-type IDH
  Participants
    IDH1 mutation | 2
    IDH 2 mutation | 0
    IDH1/2 non mutated | 34
    not determined | 13
ECOG performance status [Count of Participants; unit: Participants] — The scale was developed by the Eastern Cooperative Oncology Group (ECOG). It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 (fully independent), 1 (Restricted in physically strenuous activity but ambulatory ), 2 (Ambulatory and capable of all selfcare but unable to carry out any work activities), 3 (Capable of only limited selfcare), 4 (Completely disabled) to 5 (death).
  Participants
    score 0 | 5
    score 1 | 32
    score 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at Six Months (PFS6m)
Description: Percentage of patients who have progressed / no progress after 6 months of treatment in each of the two cohorts.
Time Frame: Baseline and after 6 months
Population: Patients were analyzed stratified by cohorts according to their EGFR mutational status: Cohort A included patients with EGFR gene amplification without EGFRvIII mutation. Cohort B included patients with EGFR gene amplification and EGFRvIII mutation.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 47
Participants
  Cohort A: number analyzed (Participants) | 30
  Cohort A: Event (PFS previous to 6 months) | 26
  Cohort A: No event | 4
  Cohort B: number analyzed (Participants) | 17
  Cohort B: Event (PFS previous to 6 months) | 16
  Cohort B: No event | 1

2. Secondary Outcome: Safety and Tolerability of Oral Administration of PF-00299804.
Description: Type, incidence, severity, frequency, severity and relationship with IMP of reported adverse events, physical examinations and laboratory tests. Toxicity will be classified and tabulated by NCI-CTCAE v 4.0.
Time Frame: Up to 42 months
Population: Safety population. All patients that were enrolled and received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 49
Participants
  Any grade Adverse event: Yes | 47
  Any grade Adverse event: No | 2
  Grade 3 or higher Adverse envent: Yes | 20
  Grade 3 or higher Adverse envent: No | 29

3. Secondary Outcome: Anti-tumor Response
Description: According to RANO criteria. Based on neurological symptoms, doses of dexamethasone and radiological response, assessed by the PI of each center. There will be central review of MRI.
Time Frame: Baseline and every 12 weeks
Population: The analisis was stratified by cohort according to their EGFR mutational status
Measure: Count of Participants; unit: Participants
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 49
Participants
  Cohort A: number analyzed (Participants) | 30
  Cohort A: Complete response | 1
  Cohort A: Partial response | 1
  Cohort A: Stable disease | 8
  Cohort A: Progressive disease | 17
  Cohort A: Not evaluable | 3
  Cohort B: number analyzed (Participants) | 19
  Cohort B: Complete response | 0
  Cohort B: Partial response | 1
  Cohort B: Stable disease | 4
  Cohort B: Progressive disease | 13
  Cohort B: Not evaluable | 1

4. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death by any cause.
Time Frame: Up to 42 months
Population: 2 patients were not evaluable because they withdrawn their consent Data is reported stratified by cohort according to their EGFR mutational status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 47
Months
  Cohort A: number analyzed (Participants) | 30
  Cohort A | 7.8 [5.6 to 10.1]
  Cohort B: number analyzed (Participants) | 17
  Cohort B | 6.7 [4.3 to 9.1]
  Full data set | 7.4 [5.6 to 9.2]

5. Secondary Outcome: Response Duration
Description: Time from first objective response up to disease progression according RANO (in patients with objective responses).
Time Frame: Baseline and every 12 weeks
Population: Data were not collected
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in the Use of Glucocorticoids
Description: Percentage of patients decreasing doses of corticosteroids during treatment.
Time Frame: Baseline and every 12 weeks
Population: Data were not collected
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in Neurological Status.
Description: By means of minimental test, it will be determined the changes in neurological status of patients.
Time Frame: Baseline and every 12 weeks
Population: Data were not collected
Arm/Group | PF-299804 (Dacomitinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period, 4 years
Description: Reported in the safety population, all patients that received at least one dose of study treatment (n= 49)
Arm/Group | PF-299804 (Dacomitinib)
All-Cause Mortality (participants affected / at risk) | 43/49
Serious Adverse Events (participants affected / at risk) | 16/49
Other Adverse Events (participants affected / at risk) | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-299804 (Dacomitinib) (N=49)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-299804 (Dacomitinib) (N=49)
Rash (Skin and subcutaneous tissue disorders) | 40
Diarrhea (Gastrointestinal disorders) | 33
Asthenia (General disorders) | 11
Vomiting (Gastrointestinal disorders) | 4

LIMITATIONS AND CAVEATS:
Important limitations of our study are the small sample size and the nonrandomized design, which preclude drawing firm conclusions, EGFR amplification, which has been used as a primary laboratory assessment, was tested in the primary tumor, and we have no evidence of the stability of this alteration in the recurrent GBs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No